CLINICAL TRIAL: NCT05920681
Title: Transanal Irrigation - Best Treatment Possibility for Low Anterior Resection Syndrome? Multicenter, Randomized Clinical Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cancer Center Affiliate of Vilnius University Hospital Santaros Klinikos (Other)
Responsible Party: Principal Investigator, Audrius Dulskas, Surgeon (oncologist), National Cancer Center Affiliate of Vilnius University Hospital Santaros Klinikos
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: LARSTAI
Record Dates: First submitted 2023-06-17; First posted 2023-06-27 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Low Anterior Resection Syndrome
Keywords: Low Anterior Resection Syndrome; Transanal irrigation; Fecal Incontinence; Colorectal Surgery; Quality of Life; Randomized Controlled Trial
MeSH Terms: conditions — Low Anterior Resection Syndrome; Fecal Incontinence

STUDY DESIGN:
Intervention Model Description: Individuals participating in this study will be randomly divided into groups 1 and 2 by randomization. The probability of falling into one or the other group is equal.
  * Group 1. This is a group of patients who will be subjected to transanal irrigation (experimental).
  * Group B. This is a group of patients who will receive only the best currently in use maintenance treatment (control).
Who Masked: Participant, Care Provider
Masking Description: During the research, the name and surname of the subject will be replaced by a special code, according to which it will not be possible to determine the identity of the subject. The subject will be randomly assigned a combination of numbers and/or letters, which will not use the patient's name, surname, initials or other personally identifiable information. This code will be used in all study documents except the consent form. If the law does not provide otherwise, only the doctor conducting the study, the research staff will be able to get acquainted with the confidential data revealing the name and surname.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transanal irrigation group (Experimental): Transanal irrigation will be applied to patients who will enter the experimental group. The patient lies on the left or right side, depending on the main hand, the knees are bent. With the main hand, he carefully introduces the TAI tip lubricated with lubricant. The TAI bag is filled with warm water - it can be boiled or just from the tap. The contents of the TAI bag are slowly administered through the anus. The duration of the TAI is about 15-20 minutes. Afterwards, the subject goes to defecate until the bowel is empty. This action should be repeated daily.
  Interventions: Procedure: Transanal irrigation
- Best supportive care group (Active Comparator): The control group will receive best supportive care (diet modification, Loperamidum if needed, diapers, etc).
  Loperamidum Dosage form: Loperamide Tablets (2mg of loperamide hydrochloride.). Dosage: Initial dose - 2 tablets immediately, then - 1 tablet after each loose stool, but not earlier than 2-3 hours after the initial dose. Do not exceed the maximum daily dose - no more than 6 tablets for adults (maximum daily dose 12 mg).
  Interventions: Combination Product: Best supportive care

INTERVENTIONS:
Procedure: Transanal irrigation — The patient lies on the left or right side, depending on the main hand, the knees are bent. With the main hand, he carefully introduces the TAI tip lubricated with lubricant. The TAI bag is filled with warm water - d it can be boiled or just from the tap. The contents of the TAI bag are slowly administered through the anus. The duration of the TAI is about 15-20 minutes. Afterwards, the subject goes to defecate until the bowel is empty. This action should be repeated daily.
  Arms: Transanal irrigation group
Combination Product: Best supportive care — Diet modification, Loperamidum if needed, diapers, etc.
  Arms: Best supportive care group

SUMMARY:
Introduction: About 50% of patients who undergo rectal resection (mostly as a treatment for rectal cancer) suffer from various and partly severe functional problems, despite the preservation of the anal fold. These complaints are summarized as low anterior resection syndrome (LARS). So far, there are no randomized clinical trials that would definitively confirm or deny the hypothesis regarding the most effective treatment for LARS.

Objectives: To evaluate whether transanal irrigation improves bowel function and quality of life in patients after rectal resection compared with the best supportive care.

Methods and analysis: Patients who have undergone low anterior resection will be approached for this study. During the patient's visit, we will assess their complaints regarding defecation problems, as well as any deterioration in their overall quality of life. To gather this information, we will have the patients fill out questionnaires such as the LARS (Low Anterior Resection Syndrome) and Wexner scale, along with quality of life questionnaires. Questionnaires and scales will be filled out again during the visit every 3 months for 1 year.

Discussion: This multicentre, randomized controlled trial will lead to a better understanding of LARS treatment. Moreover, it will be hypothesis generating and inform areas needing future prospective studies.

DETAILED DESCRIPTION:
This is a multicenter randomized clinical trial. The main objective of this clinical trial is to evaluate whether transanal irrigation improves bowel function and quality of life in patients following low anterior resection best supportive care. This will be accomplished by recording the patient's complaints (defecation, urination problems, deterioration of quality of life) after the operation, filling the LARS score (3,112), Wexner scale (123), quality of life questionnaires (EORTC CR29 (134) and Measure yourself medical outcomes profile (MYMOP)) (15) with additional questions: Would you advice this treatment to anybody else? Did your quality of live improve? Did the bowl function improve? Are you satisfied with the treatment? Did you expect the treatment would help? These questions will be rated from 0 to 5. All will be filled in again during the visit every 3 months for 12 months.

Study population All patients who developed LARS and meet the inclusion criteria will be offered participation in this clinical trial.

Recruitment Patients who have developed LARS and meet the inclusion criteria will be offered participation in this clinical trial upon consultation with an abdominal surgeon or surgeon at the National Cancer Institute clinic (or any other participating center). The patient will be given time to think as much as necessary, and all questions related to the clinical trial will be answered. The patient's decision to participate or not to participate in the study will not have any effect on his further treatment and or surveillance. Patients who have consented and signed the personal information form and the consent form will be included in the study.

Interventions During the study, transanal irrigations will be used -- which are considered safe procedures that do not pose additional risks to the patient.

TAI (Transanal irrigation):

Transanal irrigation will be applied to patients who will enter the experimental group. The patient lies on the left or right side, depending on the main hand, the knees are bent. With the main hand, he carefully introduces the TAI tip (cone catheter) lubricated with lubricant. The TAI bag is filled with warm water - d it can be boiled or just from the tap. The contents of the TAI bag are slowly administered through the anus - the cone catheter is inserted (the starting volume is 500ml of water and it evuantuale over 3-4 week period can be increased up to 1L). The duration of the TAI is about 15-20 minutes. Afterwards, the subject goes to defecate until the bowel is empty. This action should be repeated daily.

The patients will be instructed by the treating physician and will be contacted within 3-4 weeks on the course of the procedure.

In case of bleeding or abdominal pain, patients were instructed to contact the caregiver. For all other questions regarding TAI, the instructor could be contacted during office hours.

Best supportive care:

The control group will receive best supportive care (: diet modification - low fiber diet and personal recommendations were given), medications (bulky-forming agents and Loperamide®Loperamidum) if needed, diapers, etc ). All patients were instructed regarding the pelvic floor muscle training (Kegel exercise).

No patients received biofeedback therapy or any other interventions such as sacral nerve stimulation or percutaneous tibial nerve stimulation.

Assessments Data collection will take place during the patient visit . Demographic and clinical examination data will be collected from the medical documentation at the research center. During the visit, the patient's complaints (defecation, deterioration of quality of life) will be recorded after the operation, LARS, Wexner scale, quality of life questionnaires will be filled during the visit. Questionnaires and scales will be filled again during the visit every 3 months for 12 months. Other tests that will be performed during the visit will be long-term follow-up tests, an integral part of the treatment, not related to the clinical trial.

Sample size

A sample size of 40 is planned (an improvement of 5 points on the LARS scale):

* 20 transanal irrigation group (experimental)
* 20 best supportive care group (control). To demonstrate a 5 points difference (with 80% certainty) between intervention group and control, 34 patients required to be included (17 in each study arm). Taking into account drop off of 20% at least 20 patients per group will be needed. The primary endpoint was LARS score analysed by unpaired t test.After the statistical analysis , after conducting the research with this sample, the results will be statistically reliable for the Lithuanian population Outcome measures The objectives of the trial are to evaluate in what proportion of patients (percentage) transanal irrigation and in what proportion of patients (percentage) the best supportive treatment reduces the symptoms of LARS score (change in absolute score). Compare the results and evaluate the statistical reliability. The secondary outcomes would be assessing the change in single LARS score's items.

ELIGIBILITY:
Inclusion Criteria:

* Subject is an adult (≥ 18 years);
* Agrees to participate in a study;
* A low anterior resection (robotic, laparoscopic or open) was performed (anastomosis up to 5-7 cm from the anocutaneous line when assessed with a finger or endo(recto)scope);
* >12 months have passed since the operation or the closure of the ileostomy (if formed);
* No anastomotic leak or stenosis (assessed clinically, during examination, and/or proctogram);
* LARS >30 points (major LARS).

Exclusion Criteria:

* Tumor recurrence/progression
* Pregnancy
* Diagnosed with inflammatory bowel disease (ICD codes K50-59).
* Side-to-end anastomosis
* Palliative care
* Will not be able to perform irrigation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-06-18 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients for whom transanal irrigation reduced LARS symptom scores | 1 year
  Assess the proportion of patients with transanal irrigation that reduces the symptoms of LARS.
Proportion of patients for whom best supportive treatment reduced LARS symptom scores | 1 year
  Assess the proportion of patients with best supportive care that reduces the symptoms of LARS.

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute, Vilnius, Lithuania

REFERENCES:
- [Derived] Klimovskij M, Civilka I, Aleinikov A, Aukstikalnis T, Christensen P, Dulskas A. Is transanal irrigation the best treatment possibility for low anterior resection syndrome? A multicenter, randomized clinical trial: study protocol. Front Surg. 2024 May 13;11:1384815. doi: 10.3389/fsurg.2024.1384815. eCollection 2024. PMID 38803549